CLINICAL TRIAL: NCT00693095
Title: Evaluation of Recovery From Drug-Induced Lymphopenia Using Cytomegalovirus-specific T-cell Adoptive Transfer
Acronym: ERaDICATe
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: John Sampson (Other)
Responsible Party: Sponsor-Investigator, John Sampson, Professor Neurosurgery, Duke University
Organization: Duke University (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Pro00000580; SPORE Project 3; NCT00627224 (obsolete NCT alias)
Record Dates: First submitted 2008-06-03; First posted 2008-06-06 (Estimated); Last update posted 2018-01-30 (Actual); Status verified 2018-01

CONDITIONS: Glioblastoma
Keywords: Grade IV Glioblastoma Multiforme; Newly-diagnosed; CMV positive
MeSH Terms: conditions — Glioblastoma | interventions — Sodium Chloride

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Experimental): CMV-ALT + CMV-DCs
  Interventions: Biological: CMV-ALT + CMV-DCs
- 2 (Experimental): CMV-ALT + Saline
  Interventions: Biological: CMV-ALT + Saline

INTERVENTIONS:
Biological: CMV-ALT + CMV-DCs — CMV-ALT (3 X 10e7) with CMV-DCs (2 X 10e7)
  Arms: 1
Biological: CMV-ALT + Saline — CMV-ALT (3 X 10e7) with Saline
  Arms: 2

SUMMARY:
The purpose of this research study is to learn if your own immune cells can be activated and multiplied in order to help your body fight off the tumor cells in your brain. The safety of this procedure will also be studied. This procedure, called CMV-autologous lymphocyte transfer or CMV-ALT is investigational which means that it is not approved by the US Food and Drug Administration (FDA) and is still being tested in research studies. Autologous lymphocyte transfer or ALT means that you will receive your own immune cells back (and not from another donor) as a treatment after they have been activated and grown to large numbers in a clinical lab.

It is believed that the body's immune (protection) system can attack tumor cells and kill them. Immune cells called T-lymphocytes (T-cells) can recognize special proteins on the surface of tumors as a signal to attack and fight the cancer. In most patients with advanced cancer, the immune system does not adequately destroy the tumor because the white blood cells or T-cells are not stimulated enough.

Before your T-cells can become active against tumor cells, they require strong stimulation. There are special "stimulator" cells in the body called Dendritic Cells (DCs) that can take up proteins released from cancer cells and present pieces of these proteins to T lymphocytes to create this strong stimulation. Dendritic cells taken from your blood will be "pulsed" or loaded with genetic material called RNA (ribonucleic acid), which stimulates the DC to change the RNA into a protein called pp65. This protein is produced by a common virus called Cytomegalovirus (CMV) that 70-80% of us have been exposed to in our lifetime. Recently, we have found that this virus is present in many malignant brain tumors. Brain tumors are very aggressive and, for reasons we do not yet understand, are difficult for the body to attack. The CMV virus is a target in the tumor that, if attacked by your immune systems cells, may prevent your tumor from growing. We have found that we can grow immune cells to very large numbers from the blood of people who have evidence of prior exposure to this virus. You will therefore be tested to determine if you have pre-existing antibodies to this virus in order to participate in this study.

We will use your DCs to activate and grow immune cells from your blood to large numbers in a clinical laboratory. These CMV-specific immune cells, called CMV-ALT, will be returned to your body when they have become activated. It is hoped that these cells will seek out and kill tumor cells that express the CMV viral protein and not attack normal cells. The transfer of immune cells that stimulates your immune system is called adoptive immunotherapy. We will evaluate two doses of immune cells in this study (Dose 1 and Dose 2). Depending on when you are enrolled in this study you will receive either Dose 1 or 2. The first six patients enrolled on this study will receive Dose 1 (the lower dose) and the next six patients will receive Dose 2 (the higher dose). We do not know at this time if either dose is more effective or safer to administer which is why we are testing both doses. Dose 2 will be a larger number of immune cells if the treatment is found to be safe in the first six patients treated during this study.

In this study we will also see, in some randomly selected patients, if giving an injection of the DC pulsed with pp65 RNA into the skin improves the function of the CMV-ALT treatment or not. You will receive three injections under the skin of either some of the same DC that were used to stimulate your immune cells in the clinical laboratory or three injections of saline (salt solution) under the skin starting with the infusion of the CMV-ALT. It is unknown if a DC injection will be beneficial to the immune cells or not so the responses will be compared in patients who receive DC versus saline injection with their CMV-ALT. After these three injections, blood will be collected to compare the responses between patients that received saline to those that received DC injections.

DETAILED DESCRIPTION:
Six CMV seropositive patients with newly-diagnosed GBM will be randomized to receive CMV-ALT (3 x 107/Kg) with or without vaccine with CMV-DCs (2 x 107). All patients will undergo a leukapheresis after resection for harvest of PBLs for CMV-ALT and CMV-DC generation. Patients will then receive RT and concurrent TMZ at a standard targeted dose of 75 mg/m2/d. Patients with histologically or clinically-proven progressive disease during radiation, dependent on steroid supplements above physiologic levels at time of vaccination, and are unable to tolerate TMZ will be replaced. If sufficient CMV-specific T-cells can't be expanded or ALT doesn't meet release criteria, the patient will be replaced and their cells may be used to offer them another DC vaccination study, such as ATTAC Pro00003877. Remaining patients will then receive the initial cycle of TMZ at a standard targeted dose of 200mg/m2/d for 5 days 3 + 1 weeks after completing RT and will be randomized to receive CMV-DCs or saline simultaneous with CMV-ALT as vaccine #1. While the standard targeted dose of 200mg/m2/d for 5 days TMZ treatment is recommended, TMZ regimen may be adjusted at the discretion of the treating neuro-oncologist. Patients with MRI changes consistent with pseudoprogression who continue on TMZ will receive CMV-ALT with vaccinations as scheduled. Peripheral blood will be drawn at 0 hours, 24 hours, 48 hours, 72 hours, and 1 week post vaccine #1 for T-cell kinetics. DCs or saline will be given intradermally and divided equally to both inguinal regions. Vaccines #2 and #3 will occur at 2 week intervals. All patients will then undergo leukapheresis again for immunologic monitoring with specific assessment of baseline antigen-specific cellular and humoral immune responses.

If the initial dose of CMV-ALT is safe and the combination of CMV-DCs is safe and does not produce an inferior CMV pp65-specific immune response, a 3rd cohort of patients will be enrolled and receive a higher dose of CMV-ALT (3 x 108/Kg) along with vaccine with CMV-DCs (2 x 107). If the combination is unsafe or inferior only the CMV-ALT will be given. If CMV-ALT (3 x 108/Kg) is safe a 4th cohort of 3 patients will be enrolled and receive the same treatment as the 3rd cohort except the T-cells will be labeled with 111In and cultured ex vivo with 13C-glucose and their proliferation, persistence, and migration followed by peripheral blood sampling, Single Photon Emission Computed Tomography (SPECT ), and MRI.

After the initial 3 vaccines, patients will then receive subsequent TMZ cycles every 4 weeks for at least 6 cycles and up to 12 cycles after RT. TMZ will be given on days 1-5 of a 28 day cycle. Patients will then be imaged bimonthly and followed until death. This study will be halted if any 2 patients in any cohort of 3 experience a drug-related Grade IV or irreversible Grade III toxicity.

As part of standard care for these patients, upon tumor progression, participants may undergo stereotactic biopsy or resection. As this is not a research procedure consent will be obtained separately. However, if tissue is obtained, it will be used to confirm tumor progression histologically and to assess immunologic cell infiltration and pp65 antigen escape at the tumor site. Patients consenting to biopsy or resection will also be offered intratumoral vaccination with CMVpp65 LAMP-loaded, 111In-labeled DCs at the time of surgery to determine if they migrate to cervical lymph nodes.

ELIGIBILITY:
Inclusion Criteria:

* Age >18 years of age.
* GBM (WHO Grade IV) with definitive resection <4 weeks prior to leukapheresis with residual radiographic contrast enhancement on post-resection CT or MRI of <1 cm in maximal diameter in any axial plane.
* Karnofsky Performance Status (KPS ) of > 80% and a Curran Group status of I-IV.

Exclusion Criteria:

* Radiographic or cytologic evidence of leptomeningeal or multicentric disease at any time prior to vaccination.
* Prior conventional anti-tumor therapy other than steroids, RT, or TMZ.
* Pregnant or need to breast feed during the study period (Negative b-HCG test required).
* Requirement for continuous corticosteroids above physiologic levels at time of first vaccination.
* Active infection requiring treatment or an unexplained febrile (> 101.5o F) illness.
* Known immunosuppressive disease or human immunodeficiency virus infection.
* Patients with unstable or severe intercurrent medical conditions such as severe heart or lung disease.
* Allergic or unable to tolerate TMZ for reasons other than lymphopenia.
* Patients with previous inguinal lymph node dissection.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 23 (Actual)
Dates: Start 2008-09; Primary Completion 2013-12 (Actual); Study Completion 2015-04 (Actual)

PRIMARY OUTCOMES:
To evaluate if vaccinating adult patients with newly-diagnosed GBMs using CMV-DCs during recovery from therapeutic TMZ-induced lymphopenia with ALT in patients that are seropositive for CMV enhances the T-cell response. | 4 months after enrollment

SECONDARY OUTCOMES:
To evaluate the safety of ALT with CMV pp65-activated T-cells in adult patients with newly-diagnosed GBMs during recovery from therapeutic TMZ-induced lymphopenia. | 4 months from time of enrollment

CONTACTS AND LOCATIONS:
Overall Officials: Gordana Vlahovic, MD, Principal Investigator — Duke University
Locations (1):
- Duke University Medical Center, Durham, North Carolina, United States

REFERENCES:
- [Background] Reap EA, Suryadevara CM, Batich KA, Sanchez-Perez L, Archer GE, Schmittling RJ, Norberg PK, Herndon JE 2nd, Healy P, Congdon KL, Gedeon PC, Campbell OC, Swartz AM, Riccione KA, Yi JS, Hossain-Ibrahim MK, Saraswathula A, Nair SK, Dunn-Pirio AM, Broome TM, Weinhold KJ, Desjardins A, Vlahovic G, McLendon RE, Friedman AH, Friedman HS, Bigner DD, Fecci PE, Mitchell DA, Sampson JH. Dendritic Cells Enhance Polyfunctionality of Adoptively Transferred T Cells That Target Cytomegalovirus in Glioblastoma. Cancer Res. 2018 Jan 1;78(1):256-264. doi: 10.1158/0008-5472.CAN-17-0469. Epub 2017 Nov 1. PMID 29093005
- See also: Brain Tumor Center of Duke University Medical Center — http://www.cancer.duke.edu/btc/